CLINICAL TRIAL: NCT01764425
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Determine the Safety, Tolerability, Pharmacokinetics, Food Effect and Pharmacodynamics of Single and Multiple Ascending Doses of P7435 in Healthy, Overweight and/or Obese Subjects
Brief Title: Clinical Trial to Study the Safety Tolerability, Pharmacokinetics, Food Effect & Pharmacodynamics of a New Compound P7435 in Healthy, Overweight and/or Obese Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P7435/66/11
Record Dates: First submitted 2012-12-20; First posted 2013-01-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Healthy, Overweight and/or Obese Subjects
Keywords: P7435; Healthy,overweight and or obese subjects; Single ascending dose; Multiple ascending dose; Pharmacokinetics
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P7435 (Active Comparator): Tablets for once daily oral administration, For SAD part of the study dose would be 10 mg for Cohort 1; Cohorts 2, 3, 4 and 5 will be dosed subsequently at 30 mg, 100 mg, 300 mg, 1000 mg respectively Dose for MAD and food effects part of the study would be based on SAD study results
  Interventions: Drug: P7435
- Placebo (Placebo Comparator): Placebo tablets for oral administration
  Interventions: Drug: P7435

INTERVENTIONS:
Drug: P7435 — It is oral DGATI inhibitor with potential in dyslipidemia and T2DM

SUMMARY:
Clinical trial to study the safety tolerability, pharmacokinetics, food effect and pharmacodynamics of a new compound P7435 in in healthy, overweight and/or obese subjects

DETAILED DESCRIPTION:
* A phase I, randomized, double-blind, placebo-controlled, dose escalating study of P7435 to determine the safety, tolerability, pharmacokinetics, food effect and pharmacodynamics of single and multiple ascending doses of P7435.
* Subjects participating will be either healthy subjects or healthy overweight and/or obese subjects. In this study, overweight/obese are defined as subjects having a BMI of 23 kg/m2 and above.
* The study will be conducted in 3 parts as follows: Part A will consist of the Single Ascending Dose (SAD) study, Part B will consist of the Multiple Ascending Dose (MAD) study and Part C will consist of the Food Effect study.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and are able to provide a written informed consent to participate in the study.
* Healthy adult male subjects aged between 18 and 45 (both inclusive) years old
* BMI between 19 and 23 kg/m2. Overweight (BMI between 23 and 25kg/m2) and/or obese (BMI between 25 and 35 kg/m2) but otherwise healthy subjects in PartB .
* Healthy as determined by the investigator
* Smoking less than 10 cigarettes per day and able to refrain from smoking during confinement.
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, coke, chocolate, "power drinks") and grapefruit juice to admission.

Exclusion Criteria:

* Employees of the sponsor or clinical sites.
* Female subjects.
* No past or current serious diseases of any organ will be allowed. Exceptions may be non-malignant skin diseases, childhood asthma and other conditions as per the Investigator's discretion and discussed with the Sponsor a priori. History of significant gastrointestinal disease or other significant diseases including cardiac, renal or liver impairment.
* History of sleep apnea, irregular sleep/wake cycle or working in night shifts.
* Acute disease state
* History of hypo/hyperthyroidism or repeated abnormal TSH values at screening or obesity of endocrine origin.
* History of alcoholism for more than 2 years
* Positive serology for human immunodeficiency virus (HIV-1/2) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
* Positive findings in urine drug screen / alcohol breath test.
* Participation in another clinical trial within 90 days of the first drug administration.
* Intake of more than 8-10 cups of coffee and/or tea per day and consumption of methyl xanthine-containing beverages (tea, coffee, cola drinks, chocolate) within 48 hours prior to study.
* Donation of blood (i.e. 350 ml) within 90 days before Day -1 of the first treatment period.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to Day 5
  - Number of participants with adverse events in the single and multiple ascending dose studies.
Effect of food on drug concentrations | Day 1

SECONDARY OUTCOMES:
Pharmacokinetics profile (Cmax, Tmax, and AUC) | Day 1 and Day 14
  * The PK profile will be derived from the P7435 plasma concentration data.
  * A non compartmental model will be used to analyze the plasma levels of P7435

OTHER OUTCOMES:
Change from baseline in fasting glucose, insulin, C-peptide and lipids | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Dr Madhavi Latha Kodru, Principal Investigator; Dr Dharmesh Domadia, Principal Investigator
Locations (2):
- India (2):
  - Piramal Clinical Research, Hyderabad, Andhra Pradesh
  - Veeda Clinical Research, Ahmedabad, Gujarat